CLINICAL TRIAL: NCT03801772
Title: Effects of a Metronome on Functional Outcomes in Aquatic Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aultman Health Foundation (Other)
Responsible Party: Principal Investigator, Dan Fomich, Physical Therapist Assistant, Aultman Health Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AultmanRA2018.10.AF
Record Dates: First submitted 2019-01-08; First posted 2019-01-11 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Exercise Therapy
Keywords: Aquatic Therapy; Hydrotherapy; Pool Therapy

STUDY DESIGN:
Intervention Model Description: participants are assigned to one of two or more groups in parallel for the duration of the study
Who Masked: Outcomes Assessor
Masking Description: Single Blind: one party, either the investigator or participant, is unaware of the intervention assignment; also called single-masked study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metronome (Active Comparator): This arm will be using the metronome as a pacing device during aquatic exercises.
  Interventions: Device: Metronome
- Control (No Intervention): The patients will be educated on proper performance of aquatic exercises following normal physical therapy procedures. Patients will start with 10-20 repetitions of the exercises depending on their physical ability and progressed as the patient's strength and endurance improve. Each session will last approximately 30 to 45 minutes. The BORG scale (a valid, subjective measure of perceived exertion) will be used as a monitoring device to ensure that a desired level of exercise intensity is reached. The desired level is a score between 12 and 16. The patients will be asked to rate their level of exertion at the end of each session. Intensity of the exercises will be adjusted the next session if the patient's reported level of exertion does not fall within the desired range. The pain rating and the BORG number will be recorded for both groups in the chart and flow

INTERVENTIONS:
Device: Metronome — Pacing aquatic exercises to the beats per minute of a metronome. The metronome will be adjusted to each patient's pain free exertion level. Patients will start with 10-20 repetitions of the exercises depending on their physical ability. The repetitions will be progressed as the patient's strength and endurance improve and noted in the chart and the flow sheet. The metronome will be synchronized during their second aquatic therapy treatment. The beats per minute (BPM) will be increased on the metronome during the series of treatments until the patient can no longer maintain proper technique with the exercises. The exercises will continue at this BPM during future visits. The patient will be instructed to keep pace with the beat of the metronome for the duration of the exercise.
  Arms: Metronome

SUMMARY:
The purpose of this study is to determine if the use of a pacing device, a metronome, improves functional outcome measures in aquatic therapy when compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18 assigned to aquatic therapy

Exclusion Criteria:

* Women who identify themselves as pregnant on the clinics intake sheet.
* Anyone unable to hear the beats of the metronome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Change between initial 30 second sit to stand measure and final measurement | Initial evaluation and up to 8 weeks
  Patient stands and sits as many times as they can in 30 seconds. The number of repetitions is recorded.

SECONDARY OUTCOMES:
Change from the initial level reported on the Numerical Pain Rating Scale and the final reported level. | Initial evaluation and up to 8 weeks
  Pain level is reported on a 0 -10 scale with 0 being no pain and 10 being the highest level of pain.
Global Rating of Change | Up to 8 weeks
  Patient rates their improvement compared to the start of treatment from (-)7 [very much worse] to (+)7 [ completely recovered with "0" (zero) being unchanged.

CONTACTS AND LOCATIONS:
Locations (1):
- Aultman Tusc Therapy, Canton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT03801772/Prot_001.pdf